CLINICAL TRIAL: NCT04642742
Title: Impact of a Chewable Plant Sterol Supplement on LDL-C in A Real-World Setting
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Piper Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20209v4
Record Dates: First submitted 2020-11-10; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Plant sterol chewable
  Interventions: Dietary Supplement: Chewable plant sterol

INTERVENTIONS:
Dietary Supplement: Chewable plant sterol — Chewable plant sterol (gummy)

SUMMARY:
The purpose of this study is to measure the effectiveness of a twice daily plant sterol supplement, which is in a gummy format and packaged with health insights, in reducing LDL-C cholesterol in a real word setting.

DETAILED DESCRIPTION:
While the safety and benefits of plant sterol supplements have been established and are incorporated into many lipid lowering guidelines, there have been few prior studies of plant sterol chewables in gummy format among real world subjects. In this study, we aim to measure the LDL-C reducing impact of regular plant sterol supplementation in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is an adult ≥18 years of age who continuously used the sponsor's product for at least 10 weeks prior to the Follow-on Lipid Test
2. Baseline Lipid Test conducted within past 2 years
3. If smoker, smoking status or frequency has not changed between two lipid test dates
4. Subject understands the study procedures and signs forms documenting informed consent

Exclusion Criteria:

1. Subject was taking a prescription cholesterol-lowering medication or taking dietary supplements for cholesterol-lowering such as red yeast rice, niacin or omega-3 fatty acid supplements at the time of either lipid test
2. Subject does not read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Purchasers of OTC plant sterol product who have used the plant sterol product for at least 10 weeks
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-25 (Estimated); Primary Completion 2021-11-11 (Estimated); Study Completion 2021-11-11 (Estimated)

PRIMARY OUTCOMES:
% change in LDL-C from baseline | >10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Piper Biosciences, Inc., Los Altos, California, United States

IPD SHARING:
Plan to Share IPD: No